CLINICAL TRIAL: NCT07184697
Title: Efficacy and Safety of Task-specific, Biomarker-driven, High-definition, Closed-loop Transcranial Alternating Current Stimulation (HD-ctACS) in Treatment-Resistant Depression (TRD): A Randomized, Double-blind, Sham-controlled, Crossover Trial.
Brief Title: Efficacy and Safety of Task-specific, Biomarker-driven, HD-ctACS inTRD.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HD-ctACS for MDD
Record Dates: First submitted 2025-09-04; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Major Depression
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- active stimulation and crossover to sham stimulation (Active Comparator)
  Interventions: Device: HD ctACS; Device: HD ctACS sham
- sham stimulation and crossover to active stimulation (Active Comparator)
  Interventions: Device: HD ctACS; Device: HD ctACS sham

INTERVENTIONS:
Device: HD ctACS — Participants received High-Definition closed-loop transcranial Alternating Current Stimulation (HD-ctACS) for 30 minutes daily, 5 days per week. A 4x1 ring electrode montage was used, with the center electrode placed over the bilateral temporal cortices. Stimulation was delivered as a sinusoidal alternating current at a 2 mA peak amplitude, with the frequency individualized for each participant based on their baseline EEG. The stimulation was administered in a closed-loop, task-specific manner: a 500 ms burst of stimulation was triggered only when a subliminal negative facial stimulus was presented and the participant's real-time Nucleus Accumbens gamma power exceeded their baseline by two standard deviations.
Device: HD ctACS sham — Participants received High-Definition transcranial Alternating Current Stimulation (HD-tACS) in 30-minute sessions once daily, 5 days per week. A 4x1 ring electrode layout was used to target the bilateral temporal cortices. The stimulation consisted of a sinusoidal alternating current with a 2 mA peak intensity, delivered at an individualized gamma frequency determined from a baseline EEG. The intervention was administered using a closed-loop, task-specific paradigm: upon presentation of a subliminal negative facial stimulus while the real-time Nucleus Accumbens gamma power exceeded a baseline threshold of +2 SD, a 500 ms stimulation was delivered following a random delay of 1000-2000 ms.

SUMMARY:
This is a single-center, randomized, double-blind, sham-controlled, crossover exploratory clinical trial designed to evaluate the therapeutic effects of task-specific, biomarker-driven HD-ctACS on treatment-resistant depression (TRD). The study will enroll 10 patients diagnosed with TRD. Each participant will, in a randomized order, undergo a 4-week active HD-ctACS treatment period and a 4-week sham stimulation (delayed HD-ctACS) period, separated by an 8-week washout period. The primary objective is to assess the efficacy of HD-ctACS in improving core depressive symptoms, with the primary outcome being the difference in the Hamilton Depression Rating Scale (HAMD) total score between the end of the two intervention periods. Secondary objectives include evaluating the safety of the therapy, its effects on other symptom dimensions, and exploring its modulatory effects on neurobiological markers of emotional processing (e.g., NAc gamma power). The total participation time for each subject is approximately 16 weeks.

ELIGIBILITY:
Inclusion Criteria Age between 18 and 65 years, any gender.

Meets DSM-5 diagnostic criteria for Major Depressive Disorder (MDD), currently in a moderate to severe episode (total HAMD score ≥ 17).

Meets the definition of Treatment-Resistant Depression (TRD): failure to respond to or intolerance of at least two antidepressant medications from different mechanistic classes, administered at an adequate dose and duration (e.g., 6-8 weeks) during the current depressive episode.

Agrees to maintain a stable dosage of their current antidepressant medication regimen (if taking any) throughout the study period.

Able to comprehend the study procedures and voluntarily provide written informed consent.

Has intracranial deep brain electrodes implanted for research purposes, with electrodes located in the target brain regions (e.g., NAc, BNST).

Exclusion Criteria History of other severe psychiatric disorders such as schizophrenia or bipolar disorder.

Current severe suicide risk.

History of alcohol or substance abuse/dependence (within the last year).

History of epilepsy or has intracranial metal implants (other than the research electrodes).

Presence of any unstable and significant somatic illness.

Women who are pregnant or breastfeeding.

Currently participating in another clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-08-14 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Hamilton Depression Rating Scale 17-item (HAMD-17) Score | Baseline, Week 2, and Week 4 (End of Intervention).
  The 17-item Hamilton Depression Rating Scale (HAMD-17) is a clinician-rated scale used to assess the severity of depression. The total score ranges from 0 to 52. A higher score indicates a worse outcome (i.e., greater depression severity).

SECONDARY OUTCOMES:
Change from Baseline in Nucleus Accumbens (NAc) Gamma Power | Baseline, day1, day2, day3 day4, day5, day6, day7, day8, day9, day10, day11, day12, day13, day14, day15.
Amplitude of Event-Related Potential (ERP) in Response to Facial Stimuli | Baseline, day1, day2, day3 day4, day5, day6, day7, day8, day9, day10, day11, day12, day13, day14, day15.

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No